CLINICAL TRIAL: NCT01265901
Title: A Randomized, Controlled Phase III Study Investigating IMA901 Multipeptide Cancer Vaccine in Patients Receiving Sunitinib as First-line Therapy for Advanced/Metastatic Renal Cell Carcinoma
Brief Title: IMA901 in Patients Receiving Sunitinib for Advanced/Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Immatics Biotechnologies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMA901-301; 2010-022459-45 (EudraCT Number)
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-09

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic Renal Cell Carcinoma; First line; Eligible for sunitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors; sargramostim; Cyclophosphamide; IMA901 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunitinib (Active Comparator): Sunitib as Standard therapy per Label.
  Interventions: Drug: Sunitinib
- IMA901 plus GM-CSF added to sunitinib after single dose of cy (Experimental): After 1 cycle of sunitinib, intradermal vaccinations with IMA901 plus GM-CSF as adjuvant after a single dose of cyclophosphamide will be applied for a period of 4 months while continuing treatment with sunitinib
  Interventions: Drug: Sunitinib; Biological: GM-CSF; Drug: Cyclophosphamide; Drug: IMA901

INTERVENTIONS:
Drug: Sunitinib — As per label.
  Other Names: Sutent
Biological: GM-CSF — Intradermal injection of GM-CSF as adjuvant.
  Other Names: Granulocyte macrophage-colony stimulating factor; Leukine; Sargramostim
  Arms: IMA901 plus GM-CSF added to sunitinib after single dose of cy
Drug: Cyclophosphamide — One single low-dose i.v. infusion prior to the first vaccination
  Other Names: Endoxan (EU name); Cytoxan (US name)
  Arms: IMA901 plus GM-CSF added to sunitinib after single dose of cy
Drug: IMA901 — Intradermal vaccinations with IMA901 vaccine.
  Other Names: IMA901 Vaccine
  Arms: IMA901 plus GM-CSF added to sunitinib after single dose of cy

SUMMARY:
The primary objective of the phase III study is to investigate whether IMA901 can prolong overall survival in patients with metastatic and/or locally advanced renal cell carcinoma (RCC) when added to standard first-line therapy with sunitinib.

Secondary objectives include a subgroup analysis of overall survival in patients defined by a certain biomarker signature, the investigation of progression-free survival, best tumor response, safety, and immunological parameters.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized phase III study to investigate whether therapeutic vaccination with IMA901, a mult-peptide cancer vaccine (TUMAP), can prolong overall survival in patients with metastatic and/or locally advanced RCC when added to standard first-line therapy with sunitinib (primary endpoint).

Secondary endpoints include a subgroup analysis of overall survival in patients who are positive for a prospectively defined primary biomarker signature (identified as being predictive for improved clinical outcome in IMA901-vaccinated patients in the previous phase II study), progression-free survival (PFS), best overall response, cellular immunomonitoring in a subset of patients, and safety. Safety analysis will be based on adverse events (AEs), physical examinations, vital signs, hematology, clinical chemistry, urinalysis and ECG changes.

Further endpoints include subgroup analyses of overall survival in patients who are positive for further prospectively defined biomarkers (identified in the previous phase II study), and exploratory screening of new biomarkers (to be investigated in patients' blood and paraffin sections from tumor tissue) to predict better clinical outcome as response to vaccination with IMA901. Biomarker sets will not be used for patient selection in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years.
2. HLA type: HLA-A*02-positive
3. Metastatic and/or locally advanced RCC with clear cell histology (histological confirmation by local pathologist required). NOTE: prior nephrectomy is NOT required.
4. Measurable and/or non-measurable tumor lesions as per RECIST 1.1
5. Patients who are candidates for a first-line therapy with sunitinib.
6. Favorable or intermediate risk according to the 6-score risk criteria in patients treated with VEGF-targeted agents according to Heng [Heng et al. 2009]. The patient has a favorable risk if none, or intermediate risk if one or two of the following criteria apply (if three or more criteria apply the patient is not eligible):

   1. Hemoglobin < LLN,
   2. Serum corrected calcium > ULN,
   3. Karnofsky performance status < 80%,
   4. Time from initial diagnosis to initiation of therapy < 1 year,
   5. Absolute neutrophil count > ULN,
   6. Platelets > ULN.
7. Able to understand the nature of the study and give written informed consent.
8. Willingness and ability to comply with the study protocol for the duration of the study.
9. Female patients who are post menopausal (no menstrual period for a minimum of 1 year), or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) or practice a medically acceptable method of birth control.
10. Male patients willing to use contraception (upon study entry and during the course of the study or have undergone vasectomy.

Exclusion Criteria:

1. Prior systemic therapy for metastatic disease. (Note: prior adjuvant treatment for non-metastatic disease is allowed, however adjuvant therapy must have been stopped ≥ 1 year before Visit C).
2. History of or current brain metastases.
3. Abnormal ≥ CTC Grade 3 laboratory values for hematology (Hb, WBC, neutrophils, lymphocytes, platelets), liver (serum bilirubin, ALAT or ASAT) and renal function (serum creatinine).
4. Metastatic second malignancy.
5. Localized second malignancy expected to influence the patient's life span.
6. Patients with a history or evidence of systemic autoimmune disease, e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematodes (SLE), scleroderma, Sjögren's syndrome, Wegener's granulomatosis, Guillain-Barre syndrome.
7. Known active hepatitis B or C infection.
8. Known HIV infection.
9. Active infections requiring oral or intravenous antibiotics.
10. Any other known infection with a biological agent that can cause a severe disease and poses a severe danger to lab personnel working on patients' blood or tissue.
11. Received study drug within any clinical study (including approved and experimental drugs) within 4 weeks before sunitinib start.
12. Serious intercurrent illness, which according to the investigator, poses an undue risk for the patient when participating in the trial, including, but not limited to, any of the following:

    * Clinically significant cardiovascular disease (e.g., uncontrolled hypertension; clinically significant cardiac arrhythmia, clinically significant QT-prolongation),
    * New York Heart Association class III-IV congestive heart failure,
    * Symptomatic peripheral vascular disease,
    * Severe pulmonary dysfunction,
    * Psychiatric illness or social situation that would preclude study compliance.
13. Less than 12 months since any of the following:

    * Myocardial infarction,
    * Severe or unstable angina,
    * Coronary or peripheral artery bypass graft,
    * Cerebrovascular event incl. transient ischemic attack,
    * Pulmonary embolism / deep vein thrombosis (DVT).
14. Pregnancy or breastfeeding.
15. Any condition which in the judgment of the investigator would place the patient at undue risk or interfere with the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2010-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2015 (estimated)

SECONDARY OUTCOMES:
Overall survival in biomarker-defined subgroup | 2015 (estimated)
Progression-free survival | 2014 (estimated)
Best tumor response | 2014 (estimated)
Safety and tolerability | continuously
Cellular immunomonitoring | 2014 (estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rini, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute; Tim Eisen, MD, Principal Investigator — Addenbrooke's Hospital University of Cambridge, UK
Locations (105):
- United States (17):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Cedars-Siani Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Kaiser Permanente Oncology Hematology Clinic, Denver, Colorado
  - Georgetown University Medical Center, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - M.D. Anderson Cancer Center, Orlando, Florida
  - The University of Chicago Medicine, Chicago, Illinois
  - North Central Cancer Treatment Group, Illinois Cancer Care, Peoria, Illinois
  - IU Simon Cancer Center, Indianapolis, Indiana
  - Weinberg Cancer Institute at Franklin Hospital, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Clinical Research Alliance, Lake Success, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - UPMC Cancer Pavilion, University of Pittsburgh Cancer Institute, Division of Hematology / Oncology, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - South Texas Oncology & Hematology, P.A., The Start Center For Cancer Care, San Antonio, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- France (5):
  - Hôpital Saint André, Bordeaux
  - Centre Francois Baclesse, Comite Urologie-Gynecologie, Caen
  - CHU Estaing, Service d'hematologie clinique adulte et de therapie cellulaire, Clermont-Ferrand
  - Hospital Européen Georges Pompidou, Service d'oncologie medicale, Paris
  - Centre Rene Gauducheau, Service d'oncologie medicale, Saint-Herblain
- Germany (13):
  - Universitätsmedizin Berlin, Charité Campus Benjamin Franklin, Urologische Klinik und Hochschulambulanz, Berlin
  - Klinik für Hämatologie und internistische Onkologie, Augusta-Krankenanstalt gGmbH, Bochum
  - Medizinische Klinik III für Hämatologie und Onkologie, Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Essen, Klinik für Innere Medizin (Tumorforschung), Essen
  - Klinik für Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation, Medizinische Hochschule Hannover, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT), Medizinische Onkologie, Heidelberg
  - Klinik und Poliklinik für Urologie, Abteilung für Operative Medizin, Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar, Urologischen Klinik und Poliklinik, Technische Universität München, Munich
  - Urologische Klinik Dr. Castringius, München-Planegg, Planegg
  - Klinikum St. Elisabeth Straubing GmbH, Straubing
  - Klinik für Urologie, Universitätsklinikum Tübingen, Tübingen
  - Klinik für Innere Medizin III, Hämatologie - Onkologie - Rheumatologie - Infektionskrankheiten, Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen, Abteilung Hämatologie und Onkologie, Villingen-Schwenningen
- Hungary (14):
  - Péterfy Utcai Hospital, Urology department, Budapest
  - Semmelweis University, Urology Clinic, Budapest
  - Urology Department, Bajcsy-Zsilinszky Hospital, Budapest
  - Uzsoki Utcai Hospital, Oncoradiology Center, Budapest
  - University of Debrecen, Faculty of Medicine, Institute of Oncology, Debrecen
  - University of Debrecen, Faculty of Medicine, Urology Clinic, Debrecen
  - Kenézy Hospital, Urology Department, Debrecen
  - Oncology Centre, Markhot Ferenc Training Hospital and Clinic, Eger
  - Pándy Kálmán County Hospital, Oncology and Radiotherapy Center, Gyula
  - Urology department, BAZ County Hospital, Miskolc
  - Urology Clinic, University of Pécs, Pécs
  - Oncology Therapy Clinic, University of Szeged, Szeged
  - County Oncology Centre, Hetényi Géza Hospital, Szolnok
  - Oncology Department, Zala County Hospital, Zalaegerszeg
- Italy (9):
  - Presidio Ospedaliero Ospedale San Donato, U.O. Oncologia Medica, Arezzo
  - Centro di riferimento Oncologico di Aviano, Aviano
  - Medical Oncology Unit, Policlinico Sant'Orsola Malpighi, Bologna
  - Department of Oncology and Haematology, Division of Medical Oncology, University of Modena and Reggio Emilia, Modena
  - Dipartimento di Oncologia, IRCCS Fondazione, Pavia
  - Medical Oncology, Hospital Santa Maria Nuova of Reggio Emilia, Reggio Emilia
  - Oncologia Medica, "Ospedale Infermi", Rimini
  - Ospedale S.S Annunziata Sasari, Sassari
  - IRCC-Istituto di Ricerca e Cura del Cancro, Torino
- University Medical Center St. Radboud Centraal, Department of Urology, Nijmegen, Netherlands
- University Hospital, UOS - Radiumhospital, Oslo, Norway
- Poland (13):
  - Białostockie Centrum Onkologii, Bialystok
  - Prof. Franciszek Łukaszczyk Oncology Center, Bydgoszcz
  - Pomeranian Medical University Hospital, NZOZ Innowacyjna Medycyna, Dobra
  - Wojewódzki Szpital Zespolony, Oncology Department, Elblag
  - Uniwersyteckie Centrum Kliniczne, Klinika Urologii, Gdansk
  - Chemotherapy Department Center of Oncology of the Lublin Region, Lublin
  - Olsztyński Oncology Center "KOPERNIK", Olsztyn
  - Przemienienia Pańskiego Clinical Hospital no. 1, Oncology Clinic, Poznan
  - Private Outpatient Clinic MRUKMED, Rzeszów
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
  - Dzieciątka Jezus Clinical Hospital of Medical University, General Urology and Oncology Clinic, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej "Magodent", Warsaw
  - Urology and Urological Oncology Department and Clinic, Warsaw
- Romania (6):
  - Fundeni Clinical Institute, Bucharest
  - "Prof. Dr. Ioan Chiricuta" Oncology Institute, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - SC Oncolab SRL, Craiova
  - Emergency Clinical County Hospital Oradea, Oradea
  - Targu-Mures Clinical County Hospital, Oncology and Radiotherapy Department, Târgu Mureş
- Russia (17):
  - State Budget Institution of Healthcare "Chelyabinsk regional clinical oncological Dispensary", Chelyabinsk
  - Republican Clinical Oncology Dispensary of Ministry of Health of Republic Tatarstan, Kazan'
  - Institution of Russian Academy of Medical Science, "Russian Oncological Scientific Center named after N.N. Blokhin of Russian Academy of Medical Science", Moscow
  - Federal State Institution "Russian Scientific Center of Radiology and Nuclear Medicine of Healthcare of Russian Federation", Moscow
  - Moscow Hertsen Scientific Research Oncological Institute, Moscow
  - State Institution "City Clinical Hospital NO20", Moscow
  - Orenburg Regional Clinical Oncological Dispensary, Orenburg
  - State Educational Institution of High Professional Education "Rostov State Medical University of Roszdrav", Rostov-on-Don
  - State Budget Institution of Ryazan Region "Regional Clinical Oncological Diespensary", Ryazan
  - State Institution of Healthcare "Leningrad Regional Oncological Dispensary", Saint Petersburg
  - Saint-Petersburg State Institution of Healthcare "City Universal Hospital N02", Saint Petersburg
  - Saint Petersburg State Institution of Healthcare "City Clinical Oncological Dispensary", Saint Petersburg
  - Federal State Institution "Russian Scientific Center of Radiology and Surgery Technologies" of Ministry of Healthcare of Russian Federation", Saint Petersburg
  - Federal State Institution "Scientific Research Institute of Oncology named after N.N. Petrov of Ministry of Healthcare of Russian Federation", Saint Petersburg
  - Saint-Petersburg Clinical Scientific and Practical Centre of Special Methods of Medical Aid (Oncology), Saint Petersburg
  - Nonstate Institution of Healthcare "Railway clinical Hospital at Station Saratov-2 of "RZGD" PC", Saratov
  - State Institution of Healthcare of Yaroslavl Region "Regional Clinical Oncological Hospital", Yaroslavl
- United Kingdom (9):
  - Royal Bournemouth Hospital, Bournemouth
  - Addenbrooke's Hospital & Peterborough District Hospital, Cambridge University Hospitals NHS Foundation Trust, Oncology Center, Cambridge
  - Leeds Institute of Molecular Medicine, Section of Oncology and Clinical Research, St. James's University Hospital, Leeds
  - Paterson Institute for Cancer Research, Christie Hospital NHS Foundation Trust, Medical Oncology, Manchester
  - Oxford Cancer and Haematology Centre, University of Oxford, The Churchill Hospital, Oxford Radcliffe Hospital NHS Trust, Dept.of Medical Oncology, Oxford
  - ROSEMERE CANCER CENTRE, Royal Preston Hospital, Lancashire Teaching Hospital, Preston
  - CRUK Research Unit, Somers Cancer Research Building, Southampton General Hospital, Southampton
  - Postgraduate Medical School, University of Surrey, Surrey
  - South West Wales Cancer Institute, Singleton Hospital, School of Medicine, Swansea

REFERENCES:
- [Derived] Rini BI, Stenzl A, Zdrojowy R, Kogan M, Shkolnik M, Oudard S, Weikert S, Bracarda S, Crabb SJ, Bedke J, Ludwig J, Maurer D, Mendrzyk R, Wagner C, Mahr A, Fritsche J, Weinschenk T, Walter S, Kirner A, Singh-Jasuja H, Reinhardt C, Eisen T. IMA901, a multipeptide cancer vaccine, plus sunitinib versus sunitinib alone, as first-line therapy for advanced or metastatic renal cell carcinoma (IMPRINT): a multicentre, open-label, randomised, controlled, phase 3 trial. Lancet Oncol. 2016 Nov;17(11):1599-1611. doi: 10.1016/S1470-2045(16)30408-9. Epub 2016 Oct 3. PMID 27720136